CLINICAL TRIAL: NCT03730480
Title: User Performance of the CONTOUR NEXT and CONTOUR TV3 Blood Glucose Monitoring System
Brief Title: User Performance of the CONTOUR NEXT and CONTOUR TV3 Blood Glucose Monitoring System (BGMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Collaborators: Regulatory and Clinical Research Institute Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: GCA-PRO-2018-006-01
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Results first posted 2022-01-05 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects with and without Diabetes test Contour Next and Contour TV3 (Experimental): All subjects test CONTOUR NEXT BGMS and CONTOUR TV3 BGMS
  Interventions: Device: Contour Next and Contour TV3 BGMS testing by subjects with and without Diabetes

INTERVENTIONS:
Device: Contour Next and Contour TV3 BGMS testing by subjects with and without Diabetes — Using the first blood glucose monitoring system (BGMS), which is either Contour Next or Contour TV3, subjects perform self fingerstick test and alternative site test on the palm. Staff performs fingerstick test on subject. Using the second BGMS, the palm, self test and staff tests are performed. Subjects with diabetes get a venipuncture and staff tests using both BGMS using the venous blood.

SUMMARY:
This study will collect lay user ("subjects") and healthcare professional information on the performance of two different blood glucose monitors, the CONTOUR NEXT and the CONTOUR TV3, in people with and without diabetes. Each subject will use both meters, at different times and in different order, using a fingerstick(s) to collect meter samples. Meter results will be compared to standardized test system to assess the accuracy of the meters' results. Additionally, a blood sample will be drawn from the subject's arm by a trained healthcare professional for testing on both BGMS. Subjects will also be asked to complete a questionnaire to rate their experience using the meters and to evaluate the meter's Instructions for Use. After all testing and the first questionnaire have been completed, the study staff will demonstrate only to subjects with diabetes several features of the meters that would not necessarily be experienced during the meter testing. These subjects will then answer questions about the features in a second questionnaire.

DETAILED DESCRIPTION:
This clinical trial will assess the performance (accuracy) of the CONTOUR NEXT and the CONTOUR TV3 monitoring systems ("BGMS") by lay users enrolled as subjects in the study, and by health care professionals. According to a randomization schedule, subjects will be assigned to use either the CONTOUR NEXT or CONTOUR TV3 meters first and then switch and use the second meter, performing the same testing with both meters. They will learn to use the assigned meter by reading the corresponding User Guide (UG) and Quick Reference Guide (QRG). Each subject will perform one fingerstick self-test a palm (AST) test and the study staff will perform a fingerstick test on the subject. All subject self-test results and study staff results will be compared to results from the reference analyzer from a deeper fingerstick. Hematocrit will be measured for all subjects. After testing, all subjects will then complete a questionnaire (Questionnaire 1) to provide feedback on the meter system and instructions for use (UG and QRG). Subjects with diabetes will also have their glucose tested via venipuncture. After all testing is completed on these subjects, the study staff will demonstrate several features of the meter system that would not necessarily be experienced during the brief accuracy testing. These subjects with diabetes will be given a second questionnaire (Questionnaire 2) to provide feedback about the new features of the system. After completing the study procedures for one BGMS, all subjects will then repeat all of these procedures using the second BGMS, except the hematocrit and venipuncture procedures.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* Ability to speak, read and understand English. Subjects must demonstrate ability to read a paragraph from the first page of the User Guide to qualify for the study.
* Willing to complete all study procedures.

Exclusion Criteria:

* Hemophilia or any other bleeding disorder.
* Pregnancy (self-reported).
* Physical, visual or neurological impairments that would make the person unable to perform testing with the BGMS.
* Previous participation in a blood glucose monitoring study using the Ascensia CONTOUR NEXT or CONTOUR TV3 BGMS.
* Working for a medical laboratory, hospital or other clinical setting that involves training on or clinical use of blood glucose monitors.
* Working for a competitive medical device company, or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company.
* A condition, which in the opinion of the investigator or designee, would put the person or study conduct at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute; Leslie J Klaff, MD, Principal Investigator — Ranier Clinical Research Center, Inc.
Locations (2):
- United States (2):
  - AMCR Institute, Escondido, California
  - Ranier Clinical Research Center, Inc., Renton, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Persons with and without diabetes were enrolled in the study from September 06, 2018 to October 31, 2018. These subjects had one visit to the clinical trial center for the study.
Pre-assignment Details: No pre assignment
Groups:
- Contour Next and Contour TV3 -Subjects With and Without Diabetes: All subjects test CONTOUR NEXT BGMS and Contour TV3.
  Contour Next BGMS testing by subjects with and without Diabetes: All subjects perform self fingerstick test and alternative site test on the palm. Staff performs fingerstick test on subject.
  Contour TV3 BGMS: same testing as Contour Next.
  Subjects with diabetes get a venipuncture and staff tests the venous blood on both BGMS.
Period: Overall Study
Arm/Group | Contour Next and Contour TV3 -Subjects With and Without Diabetes
Started | 372
Completed | 371
Not Completed | 1
Not completed — Meter displayed a HI result which is non evaluable. | 1

BASELINE CHARACTERISTICS:
Groups:
- Contour Next BGMS and Contour TV3 BGMS -Subjects With and Without Diabetes: All subjects test CONTOUR NEXT and Contour TV3 BGMS.
  Contour Next BGMS testing by subjects with and without Diabetes: All subjects perform self fingerstick test and alternative site test on the palm. Staff performs fingerstick test on subject.
  Contour TV3 BGMS testing by subjects with and without Diabetes: All subjects perform self fingerstick test and alternative site test on the palm. Staff performs fingerstick test on subject.
  Subjects with diabetes get a venipuncture and staff tests the venous blood with both BGMS.
Arm/Group | Contour Next BGMS and Contour TV3 BGMS -Subjects With and Without Diabetes
Number analyzed (Participants) | 372
Age, Categorical [Count of Participants; unit: Participants] — age recorded per subject response Population: Some results were non evaluable due to protocol deviations, non serious AE, or no results obtained.
  Participants
    number analyzed (Participants) | 371
    <=18 years | 0
    Between 18 and 65 years | 295
    >=65 years | 76
Age, Continuous [Mean (Standard Deviation); unit: years]
  mean age | 53.1 (14.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49
  Not Hispanic or Latino | 323
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Fingerstick Contour Next BGMS and Contour TV3 Results Compared to the Reference Analyzer
Description: Number of Participants with self fingerstick results from the Contour Next BGMS and Contour TV3 BGMS that are within 15% of results from the Reference Analyzer. Results from the two meter systems will not be compared to each other.
Time Frame: 1 day
Population: Number of fingerstick self test results from Contour Next BGMS and Contour TV3 BGMS that are within 15% of reference analyzer results.
Measure: Count of Participants; unit: Participants
Groups:
- Contour Next and Contour TV3 -Subjects With and Without Diabetes: All subjects test CONTOUR NEXT BGMS and CONTOUR TV3 BGMS.
  Contour Next BGMS and Contour TV3 BGMS testing by subjects with and without Diabetes: All subjects perform self fingerstick test and alternative site test on the palm. Staff performs fingerstick test on subject. Subjects with diabetes get a venipuncture and staff tests the venous blood.
Arm/Group | Contour Next and Contour TV3 -Subjects With and Without Diabetes
Number analyzed (Participants) | 371
Participants
  Contour Next Contour Next BGMS | 366
  Contour TV3 BGMS | 360
Statistical Analysis 1: Comparison: Contour Next and Contour TV3 -Subjects With and Without Diabetes; count of number of responses; Test type: Other — count of number of results within 15% of reference analyzer; The number of results that are within 15% of reference analyzer is reported

2. Secondary Outcome: Subjects' Responses to 8 Statements Regarding Experience With Contour Next BGMS and Contour TV3 BGMS
Description: A questionnaire was given to participants with 8 statements about the BGMS instructions for use and ease of use of the meter system. These statements were rated by subjects on a Likert Scale with ratings of 1=strongly disagree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree. Participants reporting ratings greater than or equal to 3 are reported. The statements are:
  1. I find it easy to do a fingerstick blood test with this meter.
  2. The meter display is easy to see and read.
  3. It was easy to understand my test results.
  4. I like the overall meter design.
  5. I find the meter easy to use.
  6. The instructions (User Guide and Quick Reference Guide) were easy to understand.
  7. The instructions clearly explain how to run a test.
  8. The instructions clearly explain what to do if an error message is displayed by the meter.
  Note that results from the two meter systems will not be compared to each other.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Groups:
- Contour Next BGMS and Contour TV3 BGMS-Subjects With and Without Diabetes: All subjects respond to statements about CONTOUR NEXT BGMS CONTOUR TV3 BGMS.
Arm/Group | Contour Next BGMS and Contour TV3 BGMS-Subjects With and Without Diabetes
Number analyzed (Participants) | 372
Participants
  Contour Next: Responses greater than or equal to 3 for Statement 1 | 371
  Contour Next: Responses greater than or equal to 3 for Statement 2 | 371
  Contour Next: Responses greater than or equal to 3 for Statement 3 | 370
  Contour Next: Responses greater than or equal to 3 for Statement 4 | 359
  Contour Next: Responses greater than or equal to 3 for Statement 5 | 371
  Contour Next: Responses greater than or equal to 3 for Statement 6 | 367
  Contour Next: Responses greater than or equal to 3 for Statement 7 | 368
  Contour Next: Responses greater than or equal to 3 for Statement 8 | 368
  Contour TV3: Responses greater than or equal to 3 for Statement 1 | 369
  Contour TV3: Responses greater than or equal to 3 for Statement 2 | 370
  Contour TV3: Responses greater than or equal to 3 for Statement 3 | 369
  Contour TV3: Responses greater than or equal to 3 for Statement 4 | 353
  Contour TV3: Responses greater than or equal to 3 for Statement 5 | 370
  Contour TV3: Responses greater than or equal to 3 for Statement 6 | 369
  Contour TV3: Responses greater than or equal to 3 for Statement 7 | 370
  Contour TV3: Responses greater than or equal to 3 for Statement 8 | 368

ADVERSE EVENTS:
Time Frame: 1 day.
Groups:
- Contour Next BGMS and Contour TV3 BGMS -Subjects With and Without Diabetes: All subjects test CONTOUR NEXT BGMS and CONTOUR TV3 BGMS.
  Contour Next BGMS and CONTOUR TV3 BGMS testing by subjects with and without Diabetes: All subjects perform self fingerstick test and alternative site test on the palm. Staff performs fingerstick test on subject. Subjects with diabetes get a venipuncture and staff tests the venous blood.
Arm/Group | Contour Next BGMS and Contour TV3 BGMS -Subjects With and Without Diabetes
All-Cause Mortality (participants affected / at risk) | 0/372
Serious Adverse Events (participants affected / at risk) | 0/372
Other Adverse Events (participants affected / at risk) | 2/372
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contour Next BGMS and Contour TV3 BGMS -Subjects With and Without Diabetes (N=372)
Vasovagal Reaction (General disorders) | 1 (1) — The subject had a vasovagal reaction not related to the device.
Fainting (General disorders) | 1 (1) — The subject showed symptoms of fainting not related to the study device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT03730480/Prot_SAP_000.pdf